CLINICAL TRIAL: NCT02478151
Title: A Single Centre Study of the Feasibility and Safety of Using Ex-vivo Normothermic Machine Perfusion With the Organox Metra™ Device to Store Human Livers for Transplantation
Brief Title: Using Ex-vivo Normothermic Machine Perfusion With the Organox Metra™ Device to Store Human Livers for Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-8132-B
Record Dates: First submitted 2014-12-01; First posted 2015-06-23 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: End-stage Liver Disease
Keywords: Deceased donor liver transplant; Normothermic machine perfusion
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OrganOx Metra (Experimental): OrganOx Metra Device
  Interventions: Device: OrganOx Metra

INTERVENTIONS:
Device: OrganOx Metra — Normothermic machine perfusion (NMP) Metra device

SUMMARY:
This trial will examine the safety and feasibility of using the OrganOx Metra device to transport and store donor livers under normothermic conditions prior to transplantation. Participants will be followed for 3 months following transplantation and their outcomes recorded.

DETAILED DESCRIPTION:
Liver transplantation is a life-saving procedure but its success has been limited by a shortage of suitable donor organs. Much emphasis is now placed on optimising the condition of those organs that are available, to enable more higher risk organs to be transplanted safely. An effective means of pre-transplant viability assessment would not only allow greater use of higher risk donors but also minimise the risk of primary non-function by identifying and excluding non-viable organs before subjecting a patient to the risk of surgery. Organ storage under normothermic perfusion conditions enables organ function to be evaluated prior to transplantation and further has been shown to prevent organ injury which is sustained during standard cold storage. This trial will examine the safety and feasibility of using the OrganOx Metra device to transport and store donor livers under normothermic conditions prior to transplantation. This study will evaluate liver function post-transplantation using standard clinical parameters. Participants will be followed for 3 months following transplantation and their outcomes recorded. Participants will undergo no other study procedures. Feasibility will be measured using the ratio of actual / eligible candidate donors recruited to the study and will also encompass logistical issues with respect to transportation, and ease of use. Safety will be assessed by rates of device failures resulting in organ discard, primary graft non-function, re-transplantation, and recipient death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or more)
* Active on the waiting list for liver transplantation
* Able to give informed consent

Exclusion Criteria:

* Age less than 18 years
* Acute/fulminant liver failure
* Transplantation of more than one organ (e.g. liver and kidney)
* Refusal of informed consent
* Unable to give informed consent
* Re-transplantation Diagnosis of Hepatopulmonary Syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Rates of primary graft non-function | 3 months
Rates of re-transplantation | 3 months
Rates of recipient death | 3 months

SECONDARY OUTCOMES:
Rate of device failures resulting in organ discard | 3 months
Recruitment rates to the study | 3 months
  Measured by the ratio of actual / eligible candidate donors recruited to the study
Ischemia- reperfusion injury associated with organ storage | 7 days
  Assessed by a post-perfusion biopsy
Ischemia- reperfusion injury associated with organ storage | 7 days
  Assessed by measuring the peak serum aspartate transaminase level (AST) within 7 days post-transplant
The function of liver grafts stored with the Metra™ device | 3 months
  Measured by bilirubin, alkaline phosphatase, AST and INR levels at days 1-7 post-transplant. The measure is a composite.
The function of liver grafts stored with the Metra™ device | 3 months
  Measured by bilirubin, alkaline phosphatase, AST and INR levels at day 30 post-transplant. The measure is a composite.
The function of liver grafts stored with the Metra™ device | 3 months
  Measured by bilirubin, alkaline phosphatase, AST and INR levels at month 3 post-transplant. The measure is a composite.
The function of liver grafts stored with the Metra™ device | 3 months
  Measured by Lactate at days 1-3 post-transplant. The measure is a composite.
The ability of perfusion parameters to predict clinical outcomes following transplantation | 3 months
  Perfusion flows and pressures will be studied to determine their correlation with graft injury and function. The measure is a composite.
The ability of perfusion parameters to predict clinical outcomes following transplantation | 3 months
  Perfusate blood gas parameters will be studied to determine their correlation with graft injury and function. The measure is a composite.
The ability of perfusion parameters to predict clinical outcomes following transplantation | 3 months
  Bile production will be studied to determine their correlation with graft injury and function

CONTACTS AND LOCATIONS:
Overall Officials: David R Grant, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada